CLINICAL TRIAL: NCT01326533
Title: Mechanisms of Action of Hydroxychloroquine in Reducing Risk of Type 2 Diabetes
Brief Title: Reducing Risk of Type 2 Diabetes: Hydroxychloroquine Use in Pre-Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Frederico Toledo, Principal Investigator, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: DK082878; 5R21DK082878-02 (NIH)
Record Dates: First submitted 2011-03-29; First posted 2011-03-31 (Estimated); Results first posted 2016-01-29 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-01

CONDITIONS: Pre-diabetes
Keywords: pre-diabetes; hydroxychloroquine; frequently sampled intravenous glucose tolerance testing; insulin resistance; insulin secretion; glucose tolerance
MeSH Terms: conditions — Glucose Intolerance; Insulin Resistance | interventions — Hydroxychloroquine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- hydroxychloroquine (Experimental): Thirteen weeks of daily hydroxychloroquine following FSIGTT testing
  Interventions: Drug: hydroxychloroquine
- Placebo (Placebo Comparator): Thirteen weeks of daily placebo following FSIGTT testing
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: hydroxychloroquine — Thirteen weeks of oral hydroxychloroquine (400 mg/day) provided as capsules
  Other Names: Plaquenil
  Arms: hydroxychloroquine
Other: Placebo — Thirteen weeks of oral placebo provided as capsules
  Other Names: microcellulose placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the short-term effects of the antimalarial medication, hydroxychloroquine (HCQ), compared with placebo using frequently sampled intravenous glucose tolerance testing (FSIGTT) methodology to study changes in insulin secretion and glucose tolerance in subjects at risk for developing Type 2 diabetes.

DETAILED DESCRIPTION:
Diabetes is approaching epidemic proportions in the United States. This study evaluates the mechanisms of action of a generic drug that may have effects on glucose metabolism.

ELIGIBILITY:
Inclusion Criteria:

1. Age > or = 18, able to provide informed consent
2. Body-mass index greater than or equal to 25
3. Presence of at least one indicator of insulin resistance from the following list:

   * Family history of Type 2 diabetes (parent, sibling)
   * Fasting glucose 100 - 125 mg/dl
   * Fasting serum insulin greater than or equal to 7uU/ml
   * Personal history of gestational diabetes
4. Negative pregnancy test for women with childbearing potential

Exclusion Criteria:

1. Diagnosis of diabetes mellitus Type 1 or Type 2
2. Active autoimmune disease, chronic infection, current malignancy (excluding basal cell carcinoma), or other active inflammatory state that, in the opinion of the investigators, would affect insulin sensitivity
3. Oral corticosteroid use in prior six months, or expectation of needing corticosteroid therapy in upcoming six months
4. Known allergy or intolerance to HCQ
5. Known glucose-6 phosphate dehydrogenase deficiency
6. Known eye disease associated with retinal pigmentation abnormalities
7. Known diabetic retinopathy requiring past or planned laser therapy
8. Inability to comply with visit schedule and protocol requirements
9. Inability to manage and take medication as instructed
10. Current or planned pregnancy in upcoming 12 months
11. Inability or unwillingness to use reliable method of contraception (for women of childbearing years, men, or men's partners with childbearing potential), such as oral contraceptive pills, barrier method (diaphragm and condom with spermicide), intrauterine device, or depo-provera injections for 3 months prior to enrollment
12. Anemia (HGB < 9)
13. Any history of bariatric (weight loss) surgery
14. Current use of the medication Glucophage (metformin)
15. Weight changes of 6 pounds or more in the past 4 weeks
16. Any other underlying or concomitant condition, which in the opinion of the principal investigator, could confound the results of the study or put the subject at undue risk

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-03; Primary Completion 2013-03 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederico Toledo, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Montefiore Hospital, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Wasko MC, McClure CK, Kelsey SF, Huber K, Orchard T, Toledo FG. Antidiabetogenic effects of hydroxychloroquine on insulin sensitivity and beta cell function: a randomised trial. Diabetologia. 2015 Oct;58(10):2336-43. doi: 10.1007/s00125-015-3689-2. Epub 2015 Jul 22. PMID 26197707

RESULTS

PARTICIPANT FLOW:
Groups:
- Hydroxychloroquine: 13 weeks of hydroxychloroquine sulfate PO 400 mg/day
- Placebo: 13 weeks of placebo PO
Period: Overall Study
Arm/Group | Hydroxychloroquine | Placebo
Started | 17 | 15
Completed | 13 | 15
Not Completed | 4 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Hydroxychloroquine: Hydroxychloroquine sulfate PO 400 mg daily
- Placebo: Placebo daily
- Total: Total of all reporting groups
Arm/Group | Hydroxychloroquine | Placebo | Total
Number analyzed (Participants) | 17 | 15 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.1 (14.5) | 44.9 (16.8) | 47.6 (15.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 9 | 24
  Male | 2 | 6 | 8
Insulin sensitivity (Si) [Mean (Standard Deviation); unit: 10^-4 / pmol*l / min] | 0.52 (0.27) | 0.58 (0.42) | 0.55 (0.34)
Beta cell function (disposition index) [Mean (Standard Deviation); unit: arbitrary units] | 1721 (2014) | 1214 (691) | 1483 (1540)

OUTCOME MEASURES:

1. Primary Outcome: Insulin Sensitivity
Description: Change from baseline in the insulin sensitivity index (Si)
Time Frame: 13 weeks after baseline measurement
Population: all randomized with last observation carried forward for missing data
Measure: Mean (Standard Error); unit: 10^-4/pmol*l/min
Groups:
- Hydroxychloroquine: 400 mg PO daily for 13 weeks
- Placebo: PO daily for 13 weeks
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 17 | 15
10^-4/pmol*l/min | 0.08 (0.03) | -0.11 (0.04)
Statistical Analysis 1: Comparison: Hydroxychloroquine vs Placebo; Test type: Superiority or Other; p < 0.01, ANCOVA; Adjusted for baseline value as covariate

2. Secondary Outcome: Beta Cell Function
Description: Change from baseline in the disposition index (DI)
Time Frame: 13 weeks after baseline measurement
Population: all randomized with last observation carried forward for missing data
Measure: Mean (Standard Error); unit: arbitrary units
Arm/Group | Hydroxychloroquine | Placebo
Number analyzed (Participants) | 17 | 15
arbitrary units | 352 (143) | -218 (158)
Statistical Analysis 1: Comparison: Hydroxychloroquine vs Placebo; Test type: Superiority or Other; p = 0.013, ANCOVA; Adjusted for baseline value as covariate

ADVERSE EVENTS:
Time Frame: During 13 weeks of treatment
Groups:
- Hydroxychloroquine: Hydroxychloroquine sulfate PO 400mg/day
- Placebo: Placebo PO
Arm/Group | Hydroxychloroquine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/15
Other Adverse Events (participants affected / at risk) | 3/17 | 3/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydroxychloroquine (N=17) | Placebo (N=15)
Unusual or vivid dreams (General disorders) | 2 (2) | 1 (1)
Dyspepsia or GI discomfort (Gastrointestinal disorders) | 3 (3) | 3 (3)
Headache (General disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No